CLINICAL TRIAL: NCT00441129
Title: To Assess Whether Type 1 Diabetic Patients Treated With M D I and in Poor Metabolic Control Can Improve Using the Paradigm® Real Time System Compared to Self-Monitoring Blood Glucose and Continuous Subcutaneous Insulin Infusion
Brief Title: Obtain a Good Blood Glucose Control With the Paradigm Real Time System
Acronym: RTD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Diabetes (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 186
Record Dates: First submitted 2007-02-27; First posted 2007-02-28 (Estimated); Results first posted 2018-12-05 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Type 1 Diabetes
Keywords: Improvement of the blood glucose control
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional insulin pump therapy (Active Comparator): Conventional insulin pump therapy or continuous subcutaneous insulin infusion (CSII)
  Interventions: Device: Minimed Paradigm 512/712 Insulin pump
- Minimed paradigm Real Time Sytem (Experimental): Minimed paradigm Real Time Sytem
  Interventions: Device: Minimed paradigm Real Time Sytem

INTERVENTIONS:
Device: Minimed paradigm Real Time Sytem — Minimed paradigm Real Time Sytem
  Arms: Minimed paradigm Real Time Sytem
Device: Minimed Paradigm 512/712 Insulin pump — Minimed Paradigm 512/712 Insulin pump
  Arms: Conventional insulin pump therapy

SUMMARY:
In this study, subjects with insufficient metabolic control despite optimized basal-bolus injection regimens were randomily assigned to either the Mini- Med Paradigm REAL-Time insulin pump (PRT), an insulin pump that can receive and display CGM data from a separate subcutaneous glucose sensor, or conventional CSII, and compared glycemic outcomes after 6 months.

DETAILED DESCRIPTION:
The long-term clinical benefit of tight glycemic control in people with diabetes is well known . HbA1c generally assesses the average/long term quality of glycemic control, it has been clearly demonstrated that a target of HbA1c at 7.0% or less has benefits for diabetic patients

ELIGIBILITY:
Inclusion Criteria:

* Patient has signed informed consent form prior to study entry.
* Patients have been diagnosed with Type 1 DM at least 12 months prior to inclusion.
* Patients should have been received diabetes care from the investigator of each center at least 3 months prior to inclusion.
* Patients have been treated with multiple daily injections and use rapid Insulin Analog for their meal prior to study entry.
* Have an HbA1c value ≥ 8 %.
* Pediatric patients must be aged between 2 and 18 years old and adult patients be aged between 19 and 65 years old.
* Patients must perform at least 3 self-monitoring blood glucose finger-sticks daily.
* Patients from PRT group must be willing to wear sensors and transmitter connected to the pump Paradigm® Real-Time for up to 24 weeks and to change sensors, insulin infusion sets and reservoirs every 3 days (~60 times during the study period ).
* Patients from CSII group must be willing to wear an insulin pump, change insulin infusion sets, and reservoirs every 3 days (~60 times during the study period ).
* Patient is required to use the Paradigm® Real-Time system at least 70% of the time during the study period.
* Patients in both groups are required to wear at the beginning and the end of the study a CGMS for 3 days. and to perform 6 self-monitoring blood glucose finger-sticks daily during the 3 days.
* Patients must be willing to undergo all study procedures, to receive a technical training to understand how to use the Paradigm® Real-Time System or the Insulin Pump depending of the randomization.
* Patients must agree to receive a training on how to adapt their insulin doses to their meals, how to calculate and apply corrective treatment.

Exclusion Criteria:

* Hearing or vision impairment so that alarms cannot be recognized.
* Alcohol or drug abuses other than nicotine.
* Allergy to sensor or components of the sensor.
* Allergy to insulin infusion set or components of the insulin infusion set.
* Patient is pregnant or of child-bearing potential during the study.
* Patient does not have a reliable support person or the patient is unwilling to comply with the provisions of the protocol.
* Patients suffering from cancer, heart failure, kidney disease and other chronic debilitating conditions.
* Patients participating in other device or drug studies will be excluded.
* Patients may participate in this study only once.

Ages: 2 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2006-06 (Actual); Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: denis Raccah, professor, Principal Investigator — DCCT Group, Effect of Intensive Treatment of diabetes on the Development and Progression of Long-Term Complications in Insulin-Dependent Diabetes Mellitus. NJEM 1993; 329/977-986
Locations (8):
- France (8):
  - CHU Côte de Nacre, Caen
  - Hôpital Universitaire Debrousse, Lyon
  - Hôpital Sainte Marguerite, Marseille
  - CH La Peyronie, Montpellier
  - American Memorial Hospital, Reims
  - Hôpital Jeanne D'Arc, Saint-Mandé
  - Hôpitaux Universitaires de Strasbourg, Strasbourg
  - CHU Rangueil, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Raccah D, Sulmont V, Reznik Y, Guerci B, Renard E, Hanaire H, Jeandidier N, Nicolino M. Incremental value of continuous glucose monitoring when starting pump therapy in patients with poorly controlled type 1 diabetes: the RealTrend study. Diabetes Care. 2009 Dec;32(12):2245-50. doi: 10.2337/dc09-0750. Epub 2009 Sep 18. PMID 19767384

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Conventional Insulin Pump Therapy | Minimed Paradigm Real Time Sytem
Started | 60 | 55
Completed | 54 | 41
Not Completed | 6 | 14
Not completed — Withdrawal by Subject | 6 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Conventional Insulin Pump Therapy | Minimed Paradigm Real Time Sytem | Total
Number analyzed (Participants) | 60 | 55 | 115
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.8 (16.7) | 28.1 (15.1) | 28.5 (15.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 25 | 51
  Male | 34 | 30 | 64
Region of Enrollment [Number; unit: participants]
  France | 60 | 55 | 115

OUTCOME MEASURES:

1. Primary Outcome: Difference in HbA1C From Baseline and 6 Months
Description: Difference in HbA1C from Baseline and 6 Months, HbA1C at 6 months - HbA1C at baseline
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: percentage of HbA1C
Arm/Group | Conventional Insulin Pump Therapy | Minimed Paradigm Real Time Sytem
Number analyzed (Participants) | 60 | 55
percentage of HbA1C | -0.57 (0.94) | -0.81 (1.09)

2. Secondary Outcome: Change From Baseline in Mean Blood Glucose Value Calculated From CGMS Recordings.
Description: Difference in mean blood glucose value from Baseline and 6 Months, mean blood glucose value at 6 months - mean blood glucose value at baseline
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Conventional Insulin Pump Therapy | Minimed Paradigm Real Time Sytem
Number analyzed (Participants) | 60 | 55
mg/dL | -10.8 (39.6) | -30.6 (54)

3. Secondary Outcome: Change From Baseline in Total Daily Dose (TDD)
Description: Difference in TDD value from Baseline and 6 Months, TDD value at 6 months - TDD value at baseline
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: units/day
Arm/Group | Conventional Insulin Pump Therapy | Minimed Paradigm Real Time Sytem
Number analyzed (Participants) | 60 | 55
units/day | 6.8 (17.3) | 1.5 (9.1)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Conventional Insulin Pump Therapy | Minimed Paradigm Real Time Sytem
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/55
Serious Adverse Events (participants affected / at risk) | 6/60 | 2/55
Other Adverse Events (participants affected / at risk) | 25/60 | 16/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conventional Insulin Pump Therapy (N=60) | Minimed Paradigm Real Time Sytem (N=55)
Ketoacidosis (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Hypoglycemic Coma (Nervous system disorders) | 0 (0) | 1 (1)
Foot Surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Optic Neuritis (Nervous system disorders) | 1 (1) | 0 (0)
Gastroenteritis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conventional Insulin Pump Therapy (N=60) | Minimed Paradigm Real Time Sytem (N=55)
Depression (Psychiatric disorders) | 3 (3) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
Application site pain (General disorders) | 3 (3) | 0 (0)
Application site bleeding (General disorders) | 1 (1) | 0 (0)
Gastro-enteritis (Infections and infestations) | 1 (1) | 1 (1)
Sleep apnea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Abdominal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Acidoketosis (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Cutaneous irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Non-controlled diabetes mellitus (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Peripheral edema (General disorders) | 3 (3) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Visual acuity reduced (Eye disorders) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Extremity injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blindness unilateral (Eye disorders) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 3 (3) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Implantation site pruritis (General disorders) | 1 (1) | 0 (0)
Varicella (Infections and infestations) | 1 (1) | 0 (0)
Application site exfoliation (General disorders) | 1 (1) | 0 (0)
Injection site inflammation (General disorders) | 1 (1) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Allergic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Perfusion site hematoma (General disorders) | 1 (1) | 0 (0)
Hypoglycemic coma (Nervous system disorders) | 1 (1) | 0 (0)
Abcess injection site (Infections and infestations) | 1 (1) | 0 (0)
Application site erythema (General disorders) | 0 (0) | 1 (1)
Tonsilitis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Enuresis (Renal and urinary disorders) | 0 (0) | 1 (1)
Cleft lip repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Cutaneous reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Foot surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Injection site eczema (General disorders) | 0 (0) | 1 (1)
Optic neuritis (Nervous system disorders) | 0 (0) | 1 (1)
Abdominal abcess (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days